CLINICAL TRIAL: NCT04062565
Title: A Prospective Trial to Evaluate Up-front Parenteral Treprostinil and Riociguat on Right Ventriculo-vascular Coupling and Morphology in Patients With Advanced Pulmonary Arterial Hypertension (IIR-3810)
Brief Title: Trial to Evaluate Parenteral Treprostinil and Riociguat on Right Ventriculo-vascular Coupling and Morphology in Those With Advanced PAH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Franz Rischard, DO, Director, University of Arizona Pulmonary Hypertension Program, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1812168816
Record Dates: First submitted 2019-03-29; First posted 2019-08-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil; riociguat

STUDY DESIGN:
Intervention Model Description: All participants will receive Treprostinil 2-3 times per day as tolerated.
  * Subsequently, participants will receive Riociguat at 0.5 mg taken orally three times a day.
  * Participants will receive the first dose inpatient prior to discharge.
  * Participants will continue on a 2 ng/kg/min increase every other day for one week.
  * Riociguat will subsequently be increased by 0.5 mg taken orally three times a day the following week as tolerated.
  * Increases in Treprostinil and Riociguat will then alternate weeks such that only one medication is changed per week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Treprostinil and Riociguat
  Interventions: Drug: Treprostinil Injectable Product; Drug: Riociguat Pill

INTERVENTIONS:
Drug: Treprostinil Injectable Product — Injection
  Other Names: Remodulin
Drug: Riociguat Pill — Tablet
  Other Names: Adempas

SUMMARY:
The purpose of this study is to determine if there is a greater effect to patients with advanced pulmonary arterial hypertension (PAH) by using a combination of two drugs, Treprostinil and Riociquat versus Treprostinil alone

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the combined effect of parenteral treprostinil (TRE) and riociguat (RIO) versus parenteral TRE alone on right ventricular (RV)-pulmonary artery (PA) interaction (RVPA coupling) and global RV function in patients with advanced pulmonary arterial hypertension (PAH).

ELIGIBILITY:
Inclusion Criteria:

* WHO Category I PAH
* Resting mPAP ≥ 25 mmHg with a wedge pressure of ≤ 15mmHg during right heart catheterization.
* Need for parenteral TRE as determined by the PH specialist caring for the patient

Exclusion Criteria:

* Patients with a mean arterial pressure <60, and/or requiring vasopressor support
* Patients whom expected device (i.e. ECMO, RVAD) assistance or early pulmonary transplantation (within 3 months) seems inevitable
* Patients with a left ventricular ejection fraction <50% or clinical, echocardiographic, and/or catheterization data consistent with heart failure with preserved ejection fraction (HFpEF) and/or moderate-severe aortic or mitral valve abnormality
* Patients with severe restrictive lung disease (FVC<70% predicted) and/or obstructive lung disease (FEV1 <70% predicted and FEV1/FVC <70%).
* Patients with a history of pulmonary embolism within the last three months or evidence of chronic pulmonary embolism.
* Patients with a known contraindication to right heart catheterization.
* Patients whom have received active or previous pulmonary vasoactive medication within the previous 12 weeks.
* PAH associated with significant venous or capillary involvement (PCWP > 15 mmHg), known pulmonary veno-occlusive disease, and pulmonary capillary hemangiomatosis.
* Pulmonary Hypertension belonging to groups 2 to 5 of the WHO classification.
* Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C.
* Estimated creatinine clearance < 30 mL/min
* Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 1.5 times the upper limit of normal.
* Hemoglobin < 75% of the lower limit of the normal range.
* Acute or chronic physical impairment (other than dyspnea), limiting the ability to comply with study requirements.
* Pregnant or breast-feeding.

  * Females must either abstain from intercourse (when it is in line with their preferred and usual lifestyle), or
  * Use 2 medically acceptable, highly effective forms of contraception for the duration of study, and at least 30 after discontinuing study drug.
* Known concomitant life-threatening disease with a life expectancy < 12 months.
* Body weight < 40 kg and/or >150 kg.
* Any condition that prevents compliance with the protocol or adherence to therapy.
* Concurrent therapy with strong CYP3A4 inhibitors/inducers (i.e. protease inhibitors, azole antibiotics, macrolides), theophylline, and any medication in the PI's opinion may substantially potentiate the hypotensive effect of RIO.
* Treatment with nitrates of any kind within the 4 weeks prior to enrollment.
* Known hypersensitivity to drugs of the same class as TRE and/or RIO, or any of their excipients.
* Planned treatment, or treatment, with another investigational drug within 1 month prior to randomization.
* Recent (<6 months) hemoptysis and/or history of severe hemoptysis requiring intervention (bronchial artery embolization).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in stroke volume/end systolic volume (SV/ESV) | Baseline to 3 months
  Change in stroke volume/end systolic volume (SV/ESV)

SECONDARY OUTCOMES:
Change in pulmonary and cardiac pressures | Baseline to 3 months
  Increase or decrease in pressures
Change in pulmonary blood flow | Baseline to 3 months
  Increase or decrease in pulmonary blood flow
Change in end-systolic elastance/arterial elastance (Ees/Ea) | Baseline to 3 months
  Change in the interaction of the right heart and lung blood vessels
Change in Right Ventricle (RV) diastolic stiffness (Beta) | Baseline to 3 months
  Change in how stiff the wall of the right heart is at the end of relaxation
Change in 6 minute walk distance | Baseline to 3 months
  Change in how far a participant can walk during a self paced 6 minute walk test
Change in brain natriuretic peptide (BNP) | Baseline to 3 months
  Change in biomarker BNP that examines stretch on the right heart
Change in magnetic resonance imaging (MRI) right ventricle volumes | Baseline to 3 months
  Change in the volume ejected per beat and the end systolic and diastolic values of the right heart
Change in Cardio pulmonary Exercise Testing (CPET) | 3 months
  Change in how much oxygen the body consumes at peak exercise
Change in derived VO2 max | 3 months
  Change in how much oxygen the body consumes at peak exercise
Change in derived Ve/VCO2 | 3 months
  Change in how much oxygen the body consumes at peak exercise
Change in adverse event profile | Baseline to 3 months
  Change in side effects or other adverse events between combination therapy and historical control
Change in composite time to clinical worsening | Baseline to 3 months
  Difference relative to historical control in the time from diagnosis to followup, hospitalization, death or transplant

CONTACTS AND LOCATIONS:
Overall Officials: Franz Rischard, DO, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States